CLINICAL TRIAL: NCT02449291
Title: Randomised, Double-blind, Placebo-controlled Study of APD421 (Amisulpride for IV Injection) as Treatment of Established Post-operative Nausea and Vomiting, in Patients Who Have Had no Prior Prophylaxis
Brief Title: Study of APD421 as PONV Treatment (no Prior Prophylaxis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP10018
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- APD421 standard (Experimental): Single (standard) dose IV APD421
  Interventions: Drug: APD421
- APD421 high (Experimental): Single (high) dose IV APD421
  Interventions: Drug: APD421
- Placebo (Placebo Comparator): Single IV placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD421
  Arms: APD421 high; APD421 standard
Drug: Placebo
  Arms: Placebo

SUMMARY:
Double-blind, randomised, parallel-group, placebo-controlled, adaptive, seamless, dose-selecting study to compare the efficacy of APD421 to placebo as treatment of established PONV, in patients who have not had prior PONV prophylaxis.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥ 18 years of age
* Provision of written informed consent
* Patients scheduled to undergo elective surgery (open or laparoscopic technique) under general anaesthesia (other than total intravenous anaesthesia with propofol) expected to last at least one hour from induction of anaesthesia to extubation
* Patients judged by the investigator to have a low to moderate risk of experiencing PONV. In forming this judgment, investigators should pay particular attention to risk factors such as a past history of PONV and/or motion sickness; habitual non-smoking status; female sex; and likely use of opioid analgesia post-operatively
* For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (as defined in ICH M3 guidance, e.g., abstinence from sexual intercourse, surgical sterilisation (of subject or partner), combined oral contraceptive pill, a double-barrier method of contraception such as either an intra-uterine device (IUD) or an occlusive cap with spermicide, in conjunction with partner's use of a condom, or any other method or combination of methods with a failure rate generally considered to be <1% per year) between the date of screening and at least 48 hours after administration of study drug
* In order to be eligible for randomisation, subjects must also:

  (i) have experienced a first episode of PONV not more than 24 hours after the end of their operation and prior to discharge from hospital ("qualifying PONV episode"), for which they have not already received any anti-emetic treatment; and (ii) not have received any agent likely to prevent or treat nausea or vomiting (given as prophylaxis or otherwise) in the period from 12 hours prior to the start of their operation up to the time of the qualifying PONV episode.

Exclusion Criteria:

* Patients scheduled to undergo transplant surgery or any surgery where post-operative emesis may pose a significant danger to the patient
* Patients planned to receive only a local anaesthetic and/or regional neuraxial (intrathecal or epidural) block
* Patients who have received APD421 active ingredient for any indication within the last 2 weeks
* Patients who are allergic to APD421 active ingredient or any of the excipients of APD421
* Patients with a significant, ongoing history of vestibular disease or dizziness
* Patients being treated with regular anti-emetic therapy (dosed at least three times per week), which is still ongoing within one week prior to surgery
* Patients with a known prolactin-dependent tumour (e.g. pituitary gland prolactinoma or breast cancer) or phaeochromocytoma
* Patients being treated with levodopa
* Patients who are pregnant or breast feeding
* Patients with documented or suspected alcohol or substance abuse within the past 6 months
* Patients with a documented, clinically significant cardiac arrhythmia
* Patients diagnosed with Parkinson's disease
* Patients who have received emetogenic anti-cancer chemotherapy in the previous 4 weeks
* Patients with a history of epilepsy
* Any other concurrent disease or illness that, in the opinion of the investigator makes the patient unsuitable for the study
* Patients who have previously participated in this study or who have participated in another interventional clinical study involving pharmacological therapy within the previous 28 days (or longer exclusion period, if required by national or local regulations)
* Where local laws/regulations require: patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Candiotti, MD, Principal Investigator — University of Miami
Locations (4):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - Ohio State University, Columbus, Ohio
- CHU de Hautepierre, Strasbourg, France
- Universität Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Candiotti KA, Kranke P, Bergese SD, Melson TI, Motsch J, Siddiqui N, Chung F, Rodriguez Y, Minkowitz HS, Ayad SS, Diemunsch P, Fox G. Randomized, Double-Blind, Placebo-Controlled Study of Intravenous Amisulpride as Treatment of Established Postoperative Nausea and Vomiting in Patients Who Have Had No Prior Prophylaxis. Anesth Analg. 2019 Jun;128(6):1098-1105. doi: 10.1213/ANE.0000000000003733. PMID 31094774

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | APD421 Standard | APD421 High | Placebo
Started | 191 | 188 | 181
Completed | 186 | 186 | 180
Not Completed | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- APD421 5mg: APD421 5mg dose administered as a single, slow, intravenous (IV) push over about two minutes
- APD421 10mg: APD421 10mg dose administered as a single, slow, intravenous (IV) push over about two minutes
- Placebo: Matching placebo administered as a single, slow, IV push over about two minutes
- Total: Total of all reporting groups
Arm/Group | APD421 5mg | APD421 10mg | Placebo | Total
Number analyzed (Participants) | 191 | 188 | 181 | 560
Age, Continuous [Mean (Full Range); unit: years] | 44.2 [18 to 76] | 47.4 [19 to 82] | 46.5 [19 to 79] | 46.1 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 145 | 136 | 427
  Male | 45 | 43 | 45 | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 7 | 4 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 17 | 13 | 44
  White | 153 | 152 | 151 | 456
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 16 | 15 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (Success of Initial PONV Treatment)
Description: The primary efficacy variable was the dichotomous variable: success or failure of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) from 30 minutes* to 24 hours after administration of study medication and no administration of anti-emetic rescue medication at any time in the 24-hour period after administration of study medication.
Time Frame: 0-24 hours after treatment
Measure: Count of Participants; unit: Participants
Groups:
- APD421 5mg IV: APD421 (amisulpride) at 5mg administered as a single, slow, intravenous (IV) push over about two minutes.
- APD421 10mg IV: APD421 (amisulpride) at 10 mg administered as a single, slow, intravenous (IV) push over about two minutes.
- Placebo: Single IV placebo administered as a single, slow, intravenous (IV) push over about two minutes.
Arm/Group | APD421 5mg IV | APD421 10mg IV | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 60 | 59 | 39
Statistical Analysis 1: Comparison: APD421 10mg IV vs Placebo; The primary efficacy analysis was a comparison of the incidence of the primary efficacy variable between the two groups that received APD421 and the group that received placebo, using Pearson's χ2 test. The threshold for determining statistical significance in the comparison of incidence of success between the active and placebo groups (the primary efficacy analysis) was a p-value of 2.5% one-sided; Test type: Superiority; p = 0.016, Chi-squared — One-sided p-value. After adjustment for multiplicity using Hommel's method. (Note: unadjusted p value = 0.016) A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg IV vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.016, Chi-squared — One-sided p-value. After adjustment for multiplicity using Hommel's method. (Note: unadjusted p value = 0.015) A priori threshold for statistical significance = 0.025

2. Secondary Outcome: Number of Participants With Complete Response 0-2 Hrs
Description: Success of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) from 30 minutes to 2 hours after administration of study medication and no administration of anti-emetic rescue medication at any time in the 2-hour period after administration of study medication.
Time Frame: 0-2 hours after administration of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 112 | 105 | 79
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.009, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.002, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025

3. Secondary Outcome: Number of Participants With Complete Response 2-24 Hrs
Description: Success of initial PONV treatment, where success is defined as no emetic episodes (vomiting or retching) and no administration of anti-emetic rescue medication from 2 to 24 hours after administration of study medication.
Time Frame: 2-24 hours after administration of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 100 | 109 | 96
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.170, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.552, Chi-squared — One-sided p-value. No adjustment for multiple comparisons. A priori threshold for statistical significance = 0.025

4. Secondary Outcome: Time to Treatment Failure
Description: Time to first violation of the criteria for complete response
Time Frame: 0-24 hours after study drug administration
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
minutes | 159 [68 to NA] — Treatment failure occurred in less than 75% of patients | 177 [53.5 to NA] — Treatment failure occurred in less than 75% of patients | 79 [34 to 383]
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.003, Regression, Cox
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p < 0.001, Regression, Cox

5. Secondary Outcome: Number of Patients Experiencing Incidence of Emesis
Description: Number of patients experiencing vomiting or retching during the time period from 30 minutes to 24 hours after administration of study medication
Time Frame: 30 mins to 24 hours after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 64 | 57 | 62
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.209, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.440, Chi-squared

6. Secondary Outcome: Number of Participants Using Rescue Medication
Description: Proportion of patients receiving pre-specified anti-emetic rescue medication at any time in the 24 hours post-treatment period
Time Frame: 0-24 hours after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 121 | 119 | 135
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.009, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.009, Chi-squared

7. Secondary Outcome: Incidence of Significant Nausea
Description: Proportion of patients with nausea score ≥4 on an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea, therefore higher value is worse outcome) during the time period from 30 minutes to 24 hours after administration of study medication.
Time Frame: 30 mins to 24 hours after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 114 | 108 | 115
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.115, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.222, Chi-squared

8. Secondary Outcome: Incidence of Nausea
Description: Proportion of patients with nausea score ≥1 on an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea, therefore higher value is worse outcome) during the time period from 30 minutes to 24 hours after administration of study medication.
Time Frame: 30 mins to 24 hours after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Participants | 151 | 148 | 143
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.474, Chi-squared
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.505, Chi-squared

9. Secondary Outcome: Maximum Severity of Nausea
Description: Highest recorded nausea score on an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea, therefore higher value is worse outcome) during the time period from 30 minutes to 24 hours after administration of study medication.
Time Frame: 30 mins to 24 hours after study drug administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
score on a scale | 4.3 (3.24) | 4.2 (3.34) | 4.7 (3.30)
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.103, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.166, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Evolution Score of Nausea (0-30 Mins)
Description: The evolution score of nausea was calculated as the area under the curve (AUC) of the nausea scores on a scale 0-10 (where 0 is no nausea and 10 is the worst nausea imaginable) obtained at four pre-planned time points: pre-dose (0-min), and 5, 15 and 30 minutes after administration of study medication, as well as any spontaneously reported episodes of nausea during the time period, plotted against time. A higher score represents a worse outcome.
Time Frame: 0-30 minutes after study drug administration
Measure: Mean (Full Range); unit: Score on a scale*min
Arm/Group | APD421 5mg | APD421 10mg | Placebo
Number analyzed (Participants) | 191 | 188 | 181
Score on a scale*min | 1440.79 [250.0 to 3450.0] | 1502.55 [250.0 to 5375.0] | 1661.25 [250.0 to 5812.5]
Statistical Analysis 1: Comparison: APD421 10mg vs Placebo; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: APD421 5mg vs Placebo; Test type: Superiority; p = 0.029, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- APD421 5 mg: Single 5 mg dose IV APD421
- APD421 10 mg: Single 10 mg dose IV APD421
Arm/Group | APD421 5 mg | APD421 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/188 | 0/181
Serious Adverse Events (participants affected / at risk) | 5/191 | 4/188 | 5/181
Other Adverse Events (participants affected / at risk) | 43/191 | 45/188 | 49/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 5 mg (N=191) | APD421 10 mg (N=188) | Placebo (N=181)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 5 mg (N=191) | APD421 10 mg (N=188) | Placebo (N=181)
Flatulence (Gastrointestinal disorders) | 24 (25) | 17 (17) | 21 (21)
Nausea (Gastrointestinal disorders) | 15 (17) | 18 (18) | 19 (22)
Constipation (Gastrointestinal disorders) | 14 (14) | 13 (13) | 16 (16)
Infusion site pain (General disorders) | 8 (8) | 13 (13) | 7 (7)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No